CLINICAL TRIAL: NCT00000706
Title: Influence of Probenecid and Quinine on the Pharmacokinetics of Azidothymidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 027; 11003 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Quinine; Probenecid; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Quinine; Probenecid; Zidovudine

INTERVENTIONS:
Drug: Quinine sulfate
Drug: Probenecid
Drug: Zidovudine

SUMMARY:
Part I studies the effect of quinine on how zidovudine (AZT) is used by the body and eliminated through the kidneys in HIV infected patients. Part II studies the effect of probenecid and quinine on the same aspects.

Because AZT leaves the bloodstream quickly, patients must take the drug frequently to keep adequate amounts in their bodies. Probenecid and quinine may slow down the rate at which AZT leaves the body. Therefore, taking these drugs along with AZT may reduce the amount of AZT needed for treatment.

DETAILED DESCRIPTION:
Because AZT leaves the bloodstream quickly, patients must take the drug frequently to keep adequate amounts in their bodies. Probenecid and quinine may slow down the rate at which AZT leaves the body. Therefore, taking these drugs along with AZT may reduce the amount of AZT needed for treatment.

In part I, four patients who are now receiving AZT at the usual dose take part in pharmacokinetic studies (how much of the drug enters the blood stream, what happens to the drug in the body, and how it leaves the body) of AZT defined after a dose while at steady state and then again after a new steady state has been reached following the addition of quinine sulfate. Part II studies the pharmacokinetics of AZT in eight patients receiving AZT at 1 of 2 doses and then at the lower dose of AZT plus probenecid with or without quinine.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* Have symptomatic HIV infection.
* Be taking zidovudine (AZT), 100 or 200 mg, 5 or 6 x/day.

Allowed:

* History of Pneumocystis carinii pneumonia (PCP).
* Advanced AIDS related complex (ARC).
* HIV antibody positive with an absolute CD4 lymphocyte count of < 200 cells/mm3 before study entry.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions are excluded:

* Glucose-6-phosphate dehydrogenase deficiency.
* Allergy to sulfa drugs, probenecid, or quinine.

Concurrent Medication:

Excluded:

- Other drugs that might influence the metabolism or renal excretion of zidovudine (AZT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Study Completion 1988-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kornhauser D, Study Chair
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kornhauser DM, Petty BG, Hendrix CW, Woods AS, Nerhood LJ, Bartlett JG, Lietman PS. Probenecid and zidovudine metabolism. Lancet. 1989 Aug 26;2(8661):473-5. doi: 10.1016/s0140-6736(89)92087-4. PMID 2570186